CLINICAL TRIAL: NCT05299645
Title: A intervenção BeT Para Reduzir as Disparidades de prevenção e assistência ao HIV em Travestis e Mulheres Transexuais Jovens no Rio de Janeiro, Brasil
Brief Title: The BeT Study Intervention to Reduce Disparities in HIV Prevention and Care
Acronym: BET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evandro Chagas National Institute of Infectious Disease (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Raquel Malaguthi de Souza, Regulatory Affairs Associate, Evandro Chagas National Institute of Infectious Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05018818000005262; 5UG3HD096914 (NIH)
Record Dates: First submitted 2021-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: AIDS and Infections; HIV Prevention; Stigma, Social; Hiv
Keywords: Transvestites; Transsexual women; Assistance; Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Social Stigma; Helping Behavior | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: With this study, it is expected to evaluate the modification associated with the BeT intervention in prevention (engagement and adherence to PrEP) and in HIV treatment (attachment to care). Clinical trials are a powerful tool for the evaluation of health interventions, whether drug or not. Through this study, it will be possible to assess the effectiveness of a digital intervention based on peer browsing in HIV prevention and care. As this is a study with only one arm, this can interfere with obtaining measurements or verifying outcomes. To minimize the possibility of bias, the assessment of outcomes will be performed by people other than those administering the intervention. In addition, we will benchmark against an outside group, with information from the Ministry of Health's national registry systems, to determine the effect of our intervention on engagement and adherence to PrEP and linkage to HIV care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 - Transvestites and young transsexual women (Experimental): Qualitative interviews
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Pilot study with digital browsers
  Other Names: Queries

SUMMARY:
Stigma prevents young transgender women from having access to HIV prevention and care services, despite the fact that these services are freely accessible to all Brazilians in the Unified Health System (ie, SUS). Levels of HIV testing and access to care for young people are uneven. The purpose of this proposal is to generate data to address stigma in the public health system and intervene to overcome the challenges of youth with the navigation of health systems. The Brilhar e Transcender (BeT) study will include young trans women, aged 18 to 24, in Rio de Janeiro, Brazil. The BeT intervention has been found to be preliminarily efficacious in a pilot study. This proposal is for a study to test the effectiveness of an intervention to improve HIV prevention and care engagement among young trans women (N=150) at risk of HIV in Brazil.

DETAILED DESCRIPTION:
Transvestites and young transsexual women in Brazil are exposed to a high risk of exposure to HIV and poor treatment of HIV infection. Brazil remains classified as a middle-income country in 2017 [1], despite the difficult political and economic climate. In 2016, there were 830,000 adults and children living with the HIV virus [2], with a 2% increase in new infections [2]. The first population-based study to assess HIV prevalence and knowledge of pre-exposure prophylaxis (PrEP) with young trans womenin Rio de Janeiro, Brazil (Transcender Study) found that 31.2% of them were infected with HIV. In this study, among young women aged 18 to 24 years, 24.2% of them were infected with HIV, a higher rate than any other study in young trans womenin the world [3, 4], and young women had three times as many unrecognized infections as adults [5]. These findings are worse than previous research suggests, that one in five transvestites or young transsexual women under the age of 25 was infected with the HIV virus [6, 7]. Even more worrisome, the young trans women in our study had had almost twice as much unprotected anal. Adverse events assessment and reporting sex in the past three months, while their perception of HIV risk was less than half. The data reflect that there is no decline in incident infections among young women and point to a need for early intervention to reduce the risk among transvestites and young transsexual women. This is a study in collaboration with the San Francisco Department of Public Health (SFDPH). All stages will be carried out in Brazil, at the National Institute of Infectious Diseases Evandro Chagas (INI)-FIOCRUZ. People (health professionals and trans people) will be referred from four services in Rio de Janeiro, Brazil, namely: INI-FIOCRUZ, Zilda Arns Family Clinic, Luiz Capriglione Diabetes and Endocrinology Institute (IEDE) and Heitor Municipal Health Center Beltron.

The study includes the collection of formative data, the evaluation of an anti-stigma campaign and an intervention study (pilot + scale-up) of HIV prevention and treatment. The expansion provides for a Type 1 hybrid design to assess the results of the exploratory implementation and examine the results of the single-arm intervention including 150 young transvestites and trans women. We will use a pre-post design to assess intervention outcomes and include an external comparison group using data extracted from the Ministry of Health to determine the effect of our intervention on engagement and adherence to PrEP and attachment to HIV care. Implementation results will also be explored with stakeholders at partner clinics, participants and key staff. In summary, formative data will be collected with 10 young young trans women to adapt a digital systems navigation and HIV prevention and care intervention to the cultural context and HIV prevention and care needs of this population group in Brazil. A highly visible and community-informed social marketing campaign will be developed and implemented to reduce anti-trans stigma at four SUS clinics in Rio de Janeiro. To measure success, pre- and post-campaign implementation interviews will be conducted with healthcare providers at the four clinics. Additionally, a pilot, phase I study will be conducted with 20 young participants to determine the preliminary effectiveness of the antistigma campaign and navigation systems intervention and demonstrate our ability to recruit young people in this population. Exit interviews will be conducted with all pilot participants (N = 20) to collect data to refine the intervention. Finally, an expansion of the pilot intervention study will be carried out, with the inclusion of another 150 participants. At this stage, all participants will receive the BeT intervention for a period of three months, in addition to standard care for HIV prevention and care. The study includes a Type 1 hybrid design study will be conducted to assess the results of the exploratory implementation and examine the results of the single-arm intervention including 150 transvestites and young trans women. We will use a pre-post design to assess intervention outcomes and include an external comparison group using data extracted from the Ministry of Health to determine the effect of our intervention on engagement and adherence to PrEP and attachment to HIV care. n total, the participants submitted to the intervention will stay in the project for one year. The initial visit will take approximately 2 hours to develop a case management plan with a team member (ARTAS plan). As part of the intervention, volunteers will be asked to participate in a baseline behavioral survey, followed by four others over one year (ie at 3, 6, 9, and 12 months). These surveys will last approximately 1 hour. During the intervention period, the volunteers will have contact with the digital browsers at least five times via WhatsApp or other social media to check the progress of the ARTAS plan and possibly more times depending on the participant's needs.

Each interaction should not last longer than an hour. In total, participants must spend 17 hours participating in the intervention, with no maximum time to adapt to the participant's needs. Recruitment for the study will feature the FIOCRUZ team of educators, composed of three members of the trans community, in addition to the possibility of peer recruitment. Both the confirmation of eligibility and the randomization process will be carried out with double verification. The inclusion visit will be carried out in person. After the consent and eligibility verification process, participants will be included in the study and will answer questionnaires administered by trained interviewers. The Shine and Transcender (BeT) intervention was based on ARTAS, an evidencebased, individual-level, multiple-session, time-limited intervention for system navigation and linkage for HIV treatment [29]. It lasts for 3 months and is composed of BeT sessions, digital interactions, asynchronous and automatic messages. Interim analysis of primary outcomes will be performed as described in Section 9.4.6, Planned Interim Analyzes. Analyzes considering HIV serological status (HIV-positive or -negative) will be performed in accordance with Section 9.4.7, Subgroup Analysis. With this study, it is expected to evaluate the modification associated with the BeT intervention in prevention (engagement and adherence to PrEP) and in HIV treatment (attachment to care). Clinical trials are a powerful tool for the evaluation of health interventions, whether drug or not. Through this study, it will be possible to assess the effectiveness of a digital intervention based on peer browsing in HIV prevention and care. As this is a study with only one arm, this can interfere with obtaining measurements or verifying outcomes. To minimize the possibility of bias, the assessment of outcomes will be performed by people other than those administering the intervention. In addition, we will benchmark against an outside group, with information from the Ministry of Health's national registry systems, to determine the effect of our intervention on engagement and adherence to PrEP and linkage to HIV care.

ELIGIBILITY:
Intervention study:

1. Provision of signed and dated informed consent form
2. Declaration of willingness to comply with all study procedures and availability during the study
3. Age between 18 and 24 years
4. Male sex designated at birth and self-reported gender identity as a transvestite, transsexual woman or other than the designated sex
5. Desire to join the BeT intervention
6. Access to a cell phone compatible with social networks (smartphone) to participate in a technology-based intervention
7. Living in Rio de Janeiro or metropolitan area

Potential participants living with HIV must meet the following criteria:

1. Documented diagnosis of HIV infection
2. No current use of HAART OR detectable CV result OR not being followed up at a health service OR having missed at least one appointment in the last six months.

Potential HIV-negative participants must meet the following criteria:

1. No current use of PrEP
2. With indication of PrEP
3. No contraindication to PrEP

Intervention (pilot + expansion): 1) impossibility of consenting or not consenting to the research, 2) female sex assigned at birth, 3) self-identification other than transvestite, transgender woman or gender identity different from the male received at birth, 4) age under 18 or over 24 years old, 5) speak only a language other than Portuguese, 6) live outside the metropolitan region of Rio de Janeiro, 7) not have a cell phone, 8) not be sexually active.

For HIV-negative volunteers, additional criteria are:

1) being on PrEP. For HIV-positive volunteers, 1) having been diagnosed with HIV for more than one year, 2) being on regular antiretroviral therapy OR having an undetectable viral load (self-report), 3) being linked to a health service OR having attended to all consultations in the last six months.

Additionally, for the expansion phase, the following will also be considered: participation in another intervention study to promote HIV prevention or care in the last year or concomitant participation in another study that prevents concomitant inclusion (co-enrollment), refusal to perform testing for HIV, and any health condition that, in the opinion of the investigator, precludes participation in the study or harms a potential participant.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — transvestites and young transsexual women
Enrollment: 150 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Engagment on HIV prevention or care (for trans women) | 10 months
  Data from these surveys will be used to verify the primary outcomes of HIV testing, PrEP adoption, and attachment to HIV care. The results of this proposal could determine the preliminary effectiveness of the intervention in ensuring that trans youth undergo frequent HIV testing, engage in PrEP use and in HIV care.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Infectologia Evandro Chagas (Fiocruz), Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jalil EM, Wilson E, Monteiro L, Varggas T, Moura I, Torres TS, Hoagland B, Cardoso SW, Ismerio Moreira R, Goncalves Veloso Dos Santos V, Grinsztejn B; BeT Team. A Peer-Led Digital Intervention to Reduce HIV Prevention and Care Disparities Among Young Brazilian Transgender Women (The BeT Study): Protocol for an Intervention Study. JMIR Res Protoc. 2023 Feb 3;12:e44157. doi: 10.2196/44157. PMID 36735296